CLINICAL TRIAL: NCT00239447
Title: Efficacy and Safety Comparison of 4-week Treatment Periods of Two Doses [5 μg (2 Actuations of 2.5 μg) and 10 μg (2 Actuations of 5 μg)] of Tiotropium Inhalation Solution Delivered by the Respimat Inhaler, Tiotropium Inhalation Powder Capsule (18μg) Delivered by the HandiHaler in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety Comparison of Tiotropium Inhalation Solution (Respimat Inhaler) and Spiriva HandiHaler in COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.249
Record Dates: First submitted 2005-10-14; First posted 2005-10-17 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium
Device: HandiHaler
Device: Respimat SMI

SUMMARY:
Non-inferiority of lung function response to Tiotropium inhalation solution compared to Spiriva HandiHaler

ELIGIBILITY:
Inclusion criteria:

* All patients had to sign an informed consent consistent with International Conference of Harmonization-Good Clinical Practice (ICH-GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions.
* All patients had to have a diagnosis of chronic obstructive pulmonary disease.
* Patients had to have relatively stable, moderate to severe airway obstruction with an forced expiratory volume in one second (FEV1) ≤ 60% of predicted normal and FEV1 ≤ 70% of forced vital capacity FVC (Visits 1 and 2).
* Male or female patients 40 years of age or older.
* Patients had to be current or ex-smokers with a smoking history of more than 10 pack-years.
* Patients had to be able to perform technically acceptable pulmonary function tests and peak expiratory flow rate (PEFR) measurements, and had to be able to maintain records (Patient Daily Diary Card) during the study period as required in the protocol.
* Patients had to be able to inhale medication in a competent manner from the Respimat inhaler, the HandiHaler and from a metered dose inhaler (MDI).

Exclusion criteria:

* Patients with significant diseases other than chronic obstructive pulmonary disease (COPD) had to be excluded. A significant disease was defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
* Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis, if the abnormality defines a significant disease as defined in exclusion criterion No. 1.
* Patients with a recent history (i.e., one year or less) of myocardial infarction.
* Patients with any cardiac arrhythmia requiring drug therapy or who had been hospitalised for heart failure within the past three years.
* Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma were allowed.
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction.
* Patients with known narrow-angle glaucoma.
* Patients with a history of asthma, allergic rhinitis or who have a total blood eosinophil count ≥600 mm3.
* Further exclusion criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131
Dates: Start 2002-11-26 (Actual); Primary Completion 2004-04-29 (Actual); Study Completion 2004-04-29 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 response determined at the end of each 4-week period of randomised treatment. | at the end of each 4-week period

SECONDARY OUTCOMES:
Tiotropium plasma concentration data and urinary excretion data | at the end of each 4-week period
Trough forced vital capacity (FVC) response | after 4 weeks
Peak response (FEV1 and FVC) | within 3 hours after first dose, after 4 weeks
FEV1 AUC 0-12h and FVC AUC 0-12h response | after 4 weeks
FEV1 AUC 0-3h and FVC AUC 0-3h response | after the first dose, after 4 weeks
Individual FEV1and FVC measurements | during study course of 28 weeks
pre-dose morning and evening peak expiratory flow rate (PEFR) | during study course of 28 weeks
Number of occasions of rescue therapy used | during study course of 28 weeks
Median time to onset of therapeutic response after first dose (FEV1) | after first dose and after 4 weeks
Number of patients with 15% response above baseline for each treatment at each time point after first dose and after 4 weeks | up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim BV/Alkmaar
Locations (11):
- United States (10):
  - Division of Pulmonary and Critical Care Medicine, Little Rock, Arkansas
  - Boehringer Ingelheim Investigational Site, San Diego, California
  - San Jose Clinical Research, San Jose, California
  - Boehringer Ingelheim Investigational Site, Stockton, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - LSU MC-Sheveport, Shreveport, Louisiana
  - Minisota Lung Center, Minneapolis, Minnesota
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Montreal Chest Institute - McGill University Health Centre, Montreal, Quebec, Canada